CLINICAL TRIAL: NCT05848687
Title: TINI 2: Total Therapy for Infants With Acute Lymphoblastic Leukemia II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanja Andrea Gruber (Other)
Collaborators: Pediatric Oncology Experimental Therapeutics Investigators' Consortium (Unknown); Amgen (Industry); Lucile Packard Foundation for Children's Health (Unknown); Kura Oncology, Inc. (Industry); United States Department of Defense (U.S. Federal Agency); Cannonball Kid's Cancer (Unknown)
Responsible Party: Sponsor-Investigator, Tanja Andrea Gruber, Faculty - Hematology/Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-68271; PEDSHEMALL0015 (Other: Stanford OnCore)
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dexamethasone; Mitoxantrone; pegaspargase; Bortezomib; Vorinostat; Mercaptopurine; Methotrexate; blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants who meet eligibility criteria will receive remission induction, induction intensification, consolidation I, reinduction block I, reinduction block II, consolidation II, and Maintenance.
  Interventions: Dexamethasone, Mitoxantrone, PEG-asparaginase, Bortezomib, Vorinostat, Mercaptopurine, Methotrexate and Vincristine, Blinatumomab, Ziftomenib
  Interventions: Drug: Dexamethasone; Drug: Mitoxantrone; Drug: PEG asparaginase; Drug: Bortezomib; Drug: Vorinostat; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Blinatumomab; Drug: Ziftomenib

INTERVENTIONS:
Drug: Dexamethasone — Given orally (PO) or naso-gastrically (NG) or intravenously (IV).
Drug: Mitoxantrone — Given IV
Drug: PEG asparaginase — Given IV
Drug: Bortezomib — Given IV
Drug: Vorinostat — Taken PO or NG
Drug: Mercaptopurine — Given PO or NG.
Drug: Methotrexate — Given IV, IM or PO
Drug: Blinatumomab — Will be administered at 15 mcg/m2/day for 28 days following induction and reinduction
Drug: Ziftomenib — 3+3 dose escalation will be done. Dose level 1 will start at 75% of the adult recommended phase two dosing which has been established in phase I studies. Based on tolerability, we will either de-escalate to 50% RP2D (dose level -1) or escalate to 100% RP2D

SUMMARY:
The purpose of this study is to improve upon the TINI study treatment. The study will test the ability of a type of immunotherapy called blinatumomab to clear persistent leukemia. Blinatumomab targets CD19 which is located on the leukemia cells outer membrane.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≤ 365 days of age at the time of diagnosis.
* Patient has newly diagnosed CD19 positive acute lymphoblastic leukemia (ALL) or acute undifferentiated leukemia. Subjects with bilineage or biphenotypic acute leukemia are eligible provided they express CD19. Patients with CD19 positive mature B-cell ALL who carry a KMT2A rearrangement are eligible.
* Limited prior therapy, including hydroxyurea for 72 hours or less, systemic glucocorticoids for one week or less, cytarabine for 72 hours or less, one dose of vincristine, and one dose of intrathecal chemotherapy.
* Written informed consent following Institutional Review Board, NCI, FDA, and OHRP Guidelines.

Exclusion Criteria:

* Patients with prior therapy, other than therapy specified in inclusion criteria.
* Patients with mature B-cell ALL that do not have a KMT2A rearrangement or patients with acute myelogenous (AML) or T-cell ALL.
* Patients with Down syndrome.
* Inability or unwillingness of legal guardian/representative to give written informed consent

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease | 5 years and 2 months
  Proportion of patients who are minimal residual disease positive at the end of Induction Intensification

SECONDARY OUTCOMES:
Ziftomenib Minimum safe and Biologically-Effective Dose in Combination with Chemotherapy | 5 years and 6 months
  To determine the estimated minimum safe and biologically-effective dose of Ziftomenib in combination with chemotherapy, on the basis of observed DLTs, MRD assessments, and pharmacokinetic studies
Event Free Survival | 8 years
  To estimate the 3-year event-free survival for subjects treated on study
Overall Survival | 8 years
  To estimate the 3-year overall survival for subjects treated on study

CONTACTS AND LOCATIONS:
Overall Officials: Tanja A Gruber, MD, PhD, Principal Investigator — Stanford University
Locations (25):
- United States (18):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Children's Hospital of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Novant Health - Hemby Children's Hospital, Charlotte, North Carolina
  - Doernbecher Children's Hospital, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - MD Anderson, Houston, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Chu De Quebec, Québec, Quebec